CLINICAL TRIAL: NCT00271388
Title: Noise Enhanced Galvanic Vestibular Stimulation in Hemispatial Neglect
Brief Title: Vestibular Stimulation to Treat Hemispatial Neglect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Device Feasibility
Other Study IDs: C3868-R
Record Dates: First submitted 2005-12-28; First posted 2005-12-30 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Hemispatial Neglect; Stroke
Keywords: Galvanic Vestibular Stimulation; Hemispatial Neglect; Stroke
MeSH Terms: conditions — Perceptual Disorders; Stroke

STUDY DESIGN:
Who Masked: Participant

ARMS (1):
- Parameter Determination (Experimental): Testing potential effects of GVS on the symptoms of neglect
  Interventions: Device: Transcutaneous current to the vestibular nerve

INTERVENTIONS:
Device: Transcutaneous current to the vestibular nerve — Delivery of randomly oscillating low level current

SUMMARY:
The purpose of the current proposal is to pilot a new and potentially improved treatment for neglect. The procedure involves the delivery of transcutaneous small-amplitude current to the vestibular nerves that lie directly below the mastoid bones.

DETAILED DESCRIPTION:
The purpose of the current proposal is to pilot a new and potentially improved treatment for neglect. The procedure involves the delivery of transcutaneous small-amplitude current to the vestibular nerves that lie directly below the mastoid bones. With the intention of boosting activity in the damaged left hemisphere, positive and negative current is delivered to the left and right mastoids respectively. While successfully used to rehabilitate gait and balance disorders, the procedure has only once been applied to neglect.

In the present investigation, we will first confirm and then optimize the conditions under which galvanic vestibular stimulation (GVS) ameliorates neglect. This in turn will justify subsequent work (in a later funding cycle) that will demonstrate the safety and efficacy of the treatment on a much larger clinical scale, and merit the construction of a miniaturized portable device.

ELIGIBILITY:
Inclusion Criteria:

* All participants must be literate in English
* Right handed
* Have corrected near-visual acuity of 20/40 or better
* Patients must also have a minimum of twelve years education
* These inclusionary criteria are based on the data of both Black, Yu, Martin, and Szalai (90) and our own studies.

  * They are intended to assure that only patients with sufficiently severe symptoms will be admitted to our study.

Exclusion Criteria:

Exclusionary criteria include:

* Homonymous hemianopia
* Presence of a severe field cut extending toward the midline on formal perimetry (however many patients who have field cuts restricted to the periphery will be able to fully perceive our stimulus displays so can be included
* Evidence of aphasia on clinical examination (crossed aphasia)
* A significant history of other neurological or psychiatric illness or drug/alcohol abuse

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2006-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Measures of Hemispatial Neglect | 30 days
  Improvement of Hemispatial neglect

CONTACTS AND LOCATIONS:
Overall Officials: William Milberg, PhD, Principal Investigator — VA Medical Center, Jamaica Plain Campus
Locations (1):
- VA Medical Center, Jamaica Plain Campus, Boston, Massachusetts, United States